CLINICAL TRIAL: NCT01140555
Title: A Pilot Study to Determine the Optimal Procedure Steps to Obtain and Maintain Bilateral Uterine Artery Occlusion Using the GYNECARE GYNOCCLUDE™ Doppler Guided Uterine Artery Occlusion Device in Women With Uterine Fibroids
Brief Title: A Pilot Study to Determine Optimal Procedure Steps to Obtain and Maintain Uterine Artery Occlusion With the D-UAO Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Further internal evaluation of the device was required.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: David Robinson, M.D., Ethicon Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300-09-007
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GYNECARE GYNOCCLUDE™ (Experimental): GYNECARE GYNOCCLUDE™ Doppler Guided Uterine Artery Occlusion Device
  Interventions: Device: GYNECARE GYNOCCLUDE™

INTERVENTIONS:
Device: GYNECARE GYNOCCLUDE™ — GYNECARE GYNOCCLUDE™ Doppler Guided Uterine Artery Occlusion Device
  Other Names: D-UAO Device

SUMMARY:
This pilot study has a sequential design involving three groups to ensure appropriate development and evaluation of the optimal procedural steps of the D-UAO device and to confirm that those steps are reproducible in the hands of multiple surgeons.

DETAILED DESCRIPTION:
1. Group 1 - beginning with the use of the current instructions for use (IFU) will have adjustments made as necessary to the D-UAO procedural steps for uterine artery occlusion confirmed by 2/3-D Power Colour Doppler ultrasound (2/3DPD).
2. Group 2 - verify that optimal D-UAO IFU procedural steps generated in Group 1 as confirmed by 2/3DPD.
3. Group 3 - verify that the optimal D-UAO procedural steps are reproducible in the hands of multiple surgeons in addition to the group 1 investigators, as confirmed by 2/3DPD.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-55 years with regular menses and at least one symptom related to uterine fibroids (for example heavy bleeding).
* Completed child-bearing.
* At least one uterine fibroid of 3 cm diameter or greater with a prevailing pathology (e.g. as opposed to adenomyosis) of fibroids determined through abdominal/transvaginal ultrasound.
* Confirmation of the ability to clearly visualise bilateral uterine arteries with 2/3DPD.
* Dominant fibroid (defined as >3cm in diameter) must be well vascularised as determined by CE-MRI (for Group 2 and 3 patients only).
* Able to tolerate the required prolonged supine position during treatment (approximately 6 hours).
* Cervix suitable for tenaculum placement as determined by pelvic exam.
* Normal Pap smear within the last 36 months.
* Agrees to participate in the study, and following review of the patient information sheet documents this agreement by signing the Ethics Committee approved informed consent.

Exclusion Criteria:

* Prior endometrial ablation, uterine artery embolization, or uterine artery ligation.
* Pregnancy (As confirmed by a urine pregnancy test at screening and immediately prior to procedure).
* One or more lower uterine segment fibroids determined through pelvic exam which in the examiner's opinion would prevent proper clamp application.
* Any known contraindications to the contrast agent to be used for the CE-MRI as determined by the study radiologist (for Group 2 and 3 patients only).
* Pelvic mass outside the uterus suggesting other disease processes.
* An intrauterine device (IUD) in place during the day of procedure.
* Hydronephrosis as determined by interpretation of a pre-procedure renal ultrasound.
* No ureteral jets observed on ultrasound prior to clamping.
* Presence of a pedunculated fibroid determined by ultrasound, hysteroscopy, or saline infused sonography or CE MRI.
* Any current acute or chronic systemic infection or localized pelvic infection, including an unresolved urinary tract infection.
* Clinical history of any thromboembolic disease.
* History of gynecologic malignancy, atypical endometrial hyperplasia, or pelvic inflammatory disease.
* Using anticoagulation therapy (except OTC treatments, e.g. aspirin), or has a known underlying bleeding disorder.
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Optimal procedural steps | 6 hrs
  Establish and verify optimal procedural steps to obtain and maintain bilateral uterine artery occlusion using the GYNECARE GYNOCCLUDE™ Doppler Guided Uterine Artery Occlusion Device (D-UAO) for 6 hours, and confirm that these optimal procedural steps are reproducible by multiple surgeons

SECONDARY OUTCOMES:
Fibroid devascularization | Baseline and 1 month post procedure
  Evaluation of the actual and percentage change in the uterine volume, dominant fibroid volume, T2 frequency, contrast enhancement index in the dominant fibroid and the number of patient with complete infarction of all fibroid tissue obtained from a comparison of the baseline and 1 month contrast enhanced MRIs.
Safety | Baseline through one month post procedure
  Incidence of patients with adverse events that result in the following: ureteral stenting, intra-operative or post operative blood transfusion, device related hospitalization >24hours, interventional treatment for fibroids within 1 month of the D-UAO procedure, DVT or PE, life threatening cardiac or respiratory arrest or other life threatening events

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, M.D., Study Director — Ethicon, Inc.
Locations (4):
- Allgemeines Krankenhaus, Abteilung für Gynäkologie und Geburtshilfe, Linz, Austria
- Frauenklinik, Universitatsklinikum Erlangen, Erlangen, Germany
- Vrije Universiteit medisch centrum (VU Medical Center), Dept of Obstetrics and Gynaecology, Amsterdam, Netherlands
- Ullevaal University Hospital, Department of Obstetrics & Gynaecology, Oslo, Norway